CLINICAL TRIAL: NCT03349840
Title: Randomised Open Label Study of Insulin Degludec Versus Insulin Glargine U100 in Ramadan
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated by the IRB and the Institutional Official after the MOPH and WCMQ audits
Sponsor: Weill Cornell Medical College in Qatar (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1192-2978
Record Dates: First submitted 2017-11-02; First posted 2017-11-22 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Type2 Diabetes
Keywords: type 2 diabetes; insulin; glargine u100; degludec; Ramadan
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Open label randomised prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin glargine U100 (Active Comparator): Intervention: half of the subjects will be randomised to insulin glargine U100 basal insulin treatment (or continued on glargine if already treated) that will be administered daily in the evening
  Interventions: Drug: Insulin Glargine
- insulin degludec U100 (Active Comparator): Intervention: half of the subjects will be randomised to insulin degludec U100 basal insulin treatment that will be administered daily in the evening
  Interventions: Drug: Insulin Degludec U100

INTERVENTIONS:
Drug: Insulin Degludec U100 — Patients on any basal insulin including insulin glargine will be randomised and converted to basal degludec insulin
  Other Names: tresiba
  Arms: insulin degludec U100
Drug: Insulin Glargine — Patients on any basal insulin including insulin glargine will be randomised and either glargine will be continued or will beconverted to basal glargine insulin
  Other Names: lantis
  Arms: Insulin glargine U100

SUMMARY:
This is a study to be performed in Qatar that will look at the comparison of glycemic control in patients with type 2 diabetes on insulin glargine U100 with insulin degludec over the Ramadan period, to determine whether better glycemic control with fewer hypoglycemic episodes can be achieved.

DETAILED DESCRIPTION:
This will be an open label randomised prospective study that will involve 280 insulin-treated patients with type 2 diabetes and who are receiving a basal insulin as part of their treatment regimen. The power calculation suggests a subject number of 250 but to account for a 10% drop out then 280 patients will be recruited competitively. To account for an estimated 30% screen failure then 400 patients will have to be screened. Of those eligible140 patients will be randomized to insulin glargine U100 and 140 patients randomised to insulin degludec: patients will be stabilised on that regimen so that the primary objective of the study to compare glycemic control for those on insulin glargine U100 compared to those on insulin degludec can be undertaken.

Insulin glargine U100 and insulin degludec will be given once daily in the evening before Ramadan, 10-20 weeks prior to the onset of Ramadan as a run in period for stabilisation, and to be given at Iftar (breaking of the fast) in the evening of Ramadan. In accord with the latest International Diabetes Federation (IDF) guidelines the dose of both the glargine U100 and insulin degludec will be reduced by 15% during Ramadan http://www.idf.org/sites/default/files/IDF-Diabetes and Ramadan (DAR)-Practical-Guidelines-Final-Low.pdf), After Ramadan basal insulin will be increased to that of the pre-Ramadan dose. In accord with the insulin degludec label guidelines (and those of insulin glargine U100), a one to one dose will be implemented if switching from a single basal injection; however, a dose reduction of 20% will be implemented if having to switch from a twice daily basal injection (including those on twice daily insulin glargine U100 randomised to once daily insulin glargine U100). Thus, for those subjects already on once daily insulin glargine U100 and randomised to insulin glargine U100 then no dose reduction will be undertaken, nor will a dose reduction be undertaken for those subjects on once daily insulin glargine U100 and randomised to insulin degludec.

Oral hypoglycemic agents will be on a stable dose that has not been altered in the preceding 12 weeks and will be continued unchanged through the study period

During the 10-20 week run in period to Ramadan fasting blood glucose will be titrated to less than 5mmol/l (90 mg/dl)and insulin dose will be increased or decreased according to the average of three previous fasting blood glucose measurements from the previous week (weekly titration). During Ramadan fasting blood glucose will be measured before Iftar (breaking of the fast) and will aim for a fasting blood glucose of 5mmol/l (90 mg/dl).

Glycosylated hemoglobine (HbA1c) measurement will be done at baseline and 2-4 weeks before Ramadan; two weeks after Ramadan and at the end of the 8 weeks study period following Ramadan

Insulin dose will be increased by 2 units for FBG 7.1-7.9 mmol/L (120-140 mg/dl), 4 units 8.0-8.9 mmol/L (141-160 mg/dl), and 6 units 9.0 mmol/L (more than 160 mg/dl) and above. Insulin dose will be decreased by 2 units for FBG 3.1-3.9 mmol/dl (55-70 mg/dl), decreased 4 units FBG <3.1 mmol/L. During Ramadan fasting blood will be measured before Iftar. Titration of insulin will be continued for the 8 weeks following Ramadan

Patients will be contacted by a diabetes educator every 2 weeks by telephone to gather the details of their glycemic control that will be discussed with the medical investigators to alter their insulin dose and to report any hypoglycaemic events - all patients will be encouraged to measure their blood glucose if a hypoglycaemic event occurs

At the end of the study patients will have the option to be converted back to their previous basal insulin before the study. However, should they wish to continue on insulin glargine U100/ then this will be available to be continued per local guidelines.

Study Visit Schedule

Visit 1 (Initial visit: 10 to 20 weeks before Ramadan) and will include:

* Consent, inclusion and exclusion criteria, Medical history
* Anthropometric measurement - Height, Weight, Waist circumference, blood pressure.
* Blood collection for CBC, routine biochemistry including creatinine (and calculated eGFR), HbA1c, full blood count (FBC), alanine aminotransferase (ALT), sodium (NA), potassiumK (25ml)
* Electrocardiograph (ECG).

Visit 2 (within 2 weeks of visit 1: 8-18 weeks before Ramadan) and will include:

* Randomisation, randomization sequence will be created by a statistician before the start of the recruitment
* Fasting plasma glucose
* Education session and instruction on the use of the insulin degludec / glargine U100 pen. Following successful education then patients will go to pharmacy to pick up their insulin degludec/glargine U100.
* Dietary education session to optimize the effect of the change to degludec/glargine U100
* Distribution of Blood glucose meters and Diaries for the patients to record the value of their blood glucose through the period of the study.

Visit 3 (telephone calls):

Telephone calls will be conducted by the assigned clinical research coordinators (CRCs) for each subject with an interval of two weeks in which the subject will be asked about their health and readings of their blood glucose levels, they will also be asked if they had any episode of hypoglycaemia or any adverse events.

Visit 4. Just prior to Ramadan:

This is likely to be within 1-2 weeks (14 day window) before Ramadan to logistically get all patients in for that blood test.

Fasting blood will be collected for glucose, FBC, Na , K , creatinine (estimated glomerular filtration rate -eGFR), ALT and HbA1c (25ml).

Visit 5 (telephone calls):

Telephone calls will be conducted by the assigned CRCs for each subject with an interval of two weeks into Ramdan in which the subject will be asked about their health, readings of their blood glucose levels, and they will also be asked if they had any episode of hypoglycaemia or any adverse events.

Visit 6 (two weeks after Ramadan) and will include:

Fasting blood collection for glucose, FBC, HbA1c , NA , K and creatinine (eGFR estimation), ALT (25ml).

This is likely to be within 1-2 weeks (14 day window) after Ramadan to logistically get all patients in for that blood test (6 weeks between HbA1c measurements).

Visit 7 (4 weeks after visit 6 (to be done over a 14 day period) and this will include:

End of study visit and determination if patient wants to continue with insulin degludec/glargine U100 or to convert back to the basal insulin that they were on before the study

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with type 2 diabetes between the age of 20-75 years who can speak and understand Arabic or English
* Female subjects with type 2 diabetes between the age of 20-75 years who can speak and understand Arabic or English
* Patients must be on any basal insulin (once daily)
* Patients must be on any basal insulin (twice daily)
* Patients on stable dose of oral antidiabetes drugs can be included (No change in the dose for the previous 12 weeks)
* Body Mass Index <40kg/m2
* Subjects who have signed informed consent form
* Patients will be fasting during Ramadan

Exclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes on a basal bolus regimen or those on premix insulin or on self-mix insulin
* On GLP-1 receptor agonists medication
* On glinide medication
* Ischaemic heart disease
* Left bundle branch block on ECG
* Active diabetic retinopathy or maculopathy requiring acute treatment
* Unwilling to follow the protocol
* Pregnancy, intention to become pregnant, breastfeeding

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the glycemic control of insulin glargine U100 with insulin degludec in patients with type 2 diabetes from baseline to end of Ramadan. | 6 weeks
  To measure HbA1c at the end of Ramadan between arms.

SECONDARY OUTCOMES:
Comparison of the glucose control of insulin glargine U100 with insulin degludec in patients with type 2 diabetes from baseline to end of Ramadan. | 6 weeks
  To measure fasting glucose at the end of Ramadan between arms.
Hypoglycemia between arms | 6 weeks
  To measure the number hypoglycemia between arms to the end of Ramadan
HbA1c end point achieved | 6 weeks
  To measure the number of subjects who achieve a HbA1c <7.5% at the end of Ramadan between treatment arms
Incidence of Treatment-Emergent Adverse Events | 14-24 weeks
  To measure the number of adverse events between the 2 treatment arms before and after Ramadan

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Atkin, MD, Principal Investigator — Weill Cornell Medicine Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data